CLINICAL TRIAL: NCT05830682
Title: Effect of Using Walking Aid on Pain and Mobility Levels of Patients Underwent CABG Surgery
Brief Title: Effect of Using Walking Aid on Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Seher Ünver, Associate Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018/235
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Bypass Graft Surgery; Pain; Early Mobilization; Walking, Difficulty
MeSH Terms: conditions — Pain; Mobility Limitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The observer and data analysed was completed by independent researchers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this study group asked to walk with using a walking aid during the first three mobilizations in the intensive care unit on the first postoperative day.
  Interventions: Device: using a walking aid
- Control Group (No Intervention): Participants in this study group asked to walk with the help of 2 nurses during the first three mobilizations in the intensive care unit on the first postoperative day.

INTERVENTIONS:
Device: using a walking aid — The walking aid utilized for mobilizing patients in the intervention group during the study is a four-wheeled device that allows for movement in all directions. The height of the device can be adjusted according to the patients' height. It features a seat for resting when needed and a braking system that is controlled from the hand grips.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of using walking aid during out-of-bed mobilization of patients who underwent open coronary artery bypass graft surgery on levels of pain and mobility. The main hypotheses are:

1. The pain level of patients using walking aid is lower than that of those who do not.
2. The mobility level of patients using walking aid is higher than that of those who do not.

Participants will be asked to walk with using a walking aid during the first three mobilizations in the intensive care unit on the first postoperative day.

DETAILED DESCRIPTION:
Group allocation of the patients was done through using Random Allocation Software program and patients were allocated into two groups: the intervention group and the control group.

Patients in the intervention group were asked to o walk with using a walking aid during the first three mobilizations in the intensive care unit on the first postoperative day.

The researcher visited the patients in the CICU on the first day after surgery informed them that they were going to be mobilized out of the bed and walk in the room for two rounds (approximately 24 meters) for three times following each 4 hours by using a walking aid. The patients in the control group were informed that they were to be mobilized out of the bed and walk in the room for two rounds (approximately 24 meters) for three times following each 4 hours with the help of two nurses.

In the intervention group, to perform the first out-of-bed mobilization, the researcher and one other nurse supported helped the patient to straightening up in bed and then to sit in the bed. Then, the patient sat on the edge of the bed with their feet dangling outside. Following, with the brakes closed on the walking aid, the patient stood up from the bed and walked two rounds in the CICU room. The patient was then helped back to sit on the edge of the bed, and was asked to mark the level of pain and difficulty experienced during each activity on a horizontal line in the patient mobility scale.

The Patient Mobility Scale scale was developed to measure the pain and difficulty levels experienced by patients during four activities (turning from one side to the other/straightening up in bed, sitting on the edge of the bed, standing up from the bed, and walking in the room) in the postoperative period. To evaluate pain, patients are asked to mark their level of pain for each activity on a line ranging from 0-"no pain" to 5-"worst pain imaginable." To evaluate difficulty, patients are asked to mark their perceived difficulty for each activity on a line ranging from 0-"very easy" to 5-"very difficult". The total score of the patient mobility scale is derived by summing the pain and difficulty scores for all activities, with the lowest possible score being 0 and the highest score being 120. A lower score signifies that patients experienced less pain and difficulty during their activities, indicating a higher mobility level.

In the control group, to perform the first out-of-bed mobilization, the researcher and one other nurse supported helped the patient to straightening up in bed and then to sit in the bed. Then, the patient sat on the edge of the bed with their feet dangling outside. Following, two nurses helped the patient stood up from the bed and walk two rounds in the CICU room. The patient was then helped back to sit on the edge of the bed and was asked to mark the level of pain and difficulty experienced during each activity on a horizontal line in the patient mobility scale.

Four hours after the first and second mobilizations, both groups of patients underwent a new mobilization procedure, and the interventions applied during the first mobilization were repeated.

ELIGIBILITY:
Inclusion Criteria:

* underwent elective CABG surgery for the first-time
* received sternotomy during surgery
* had saphenous vein grafting
* were within the first day after surgery
* being volunteered to participate in the study

Exclusion Criteria:

* patients who had a vein other than the saphenous vein grafting
* whose mobilization was not approved by the physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Pain level | in the intensive care unit on the first postoperative day
  will be evaluated with using the Patient Mobility Scale. To evaluate pain, patients are asked to mark their level of pain for each activity on a line ranging from 0-"no pain" to 5-"worst pain imaginable."
Difficulty level | in the intensive care unit on the first postoperative day
  will be evaluated with using the Patient Mobility Scale. To evaluate difficulty, patients are asked to mark their perceived difficulty for each activity on a line ranging from 0-"very easy" to 5-"very difficult"

CONTACTS AND LOCATIONS:
Overall Officials: Seher Ünver, Principal Investigator — Trakya University; Simge R Aktürk Tuncer, Principal Investigator — Çorlu State Hospital
Locations (1):
- Seher Ünver, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No